CLINICAL TRIAL: NCT07378774
Title: Constraint-Induced Movement Therapy and Bilateral Training in Chronic Stroke
Brief Title: Constraint Induced Movement Therapy and Bilateral Training in Chronic Stroke
Acronym: CIMT-BT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zikra Azhar (Other)
Responsible Party: Sponsor-Investigator, Zikra Azhar, principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/15/03/40
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Stroke
Keywords: Chronic stroke; Constraint-induced movement therapy; Bilateral training; Upper limb rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A CIMT (Experimental): Participants in this arm will receive Constraint-Induced Movement Therapy combined with Functional Electrical Stimulation (FES). The non-affected upper limb will be restrained using a mitt or glove to encourage use of the affected limb during therapy sessions. Task-oriented and functional activities focusing on grasping, releasing, reaching, and object manipulation will be practiced with the affected upper limb. Functional Electrical Stimulation will be applied to the wrist extensor muscles to facilitate muscle activation, reduce spasticity, and enhance motor recovery. Therapy will be provided three sessions per week for eight weeks.
  Interventions: Behavioral: CIMT
- group B bilateral training (Active Comparator): Participants in this arm will receive Bilateral Training combined with Functional Electrical Stimulation (FES). Therapy will involve simultaneous use of both upper limbs to perform symmetrical and functional task-based activities aimed at improving coordination and motor control of the affected limb. Tasks will progress from simple bilateral movements to functional activities involving both hands. Functional Electrical Stimulation will be applied to the wrist extensor muscles using the same parameters as the experimental group. Therapy will be delivered three sessions per week for eight weeks.
  Interventions: Behavioral: bilateral training

INTERVENTIONS:
Behavioral: CIMT — Constraint-Induced Movement Therapy (CIMT) will be administered by restraining the non-affected upper limb using a mitt or glove to promote active use of the affected limb. Participants will perform task-oriented and functional activities such as grasping, releasing, reaching, object manipulation, and activities of daily living using the affected upper limb. Training intensity will be progressively increased based on patient performance. Functional Electrical Stimulation (FES) will be applied to the wrist extensor muscles (extensor carpi radialis longus and brevis) to facilitate muscle contraction, reduce spasticity, and enhance motor relearning. Sessions will be conducted three times per week for eight weeks.
  Other Names: Constrain induced movement therapy
  Arms: group A CIMT
Behavioral: bilateral training — Bilateral Training will involve simultaneous use of both upper limbs to perform symmetrical and functional task-based activities designed to improve coordination and motor control of the affected upper limb. Exercises will progress from simple bilateral movements to complex functional tasks such as lifting objects, folding towels, and opening containers. Functional Electrical Stimulation (FES) will be applied to the wrist extensor muscles using the same stimulation parameters as the experimental intervention to ensure consistency. Therapy will be delivered three times per week for eight weeks.
  Arms: group B bilateral training

SUMMARY:
Stroke is a leading cause of long-term disability, with upper limb spasticity and impaired hand function being common problems in the chronic phase. These impairments significantly affect independence in activities of daily living and overall quality of life. Constraint-Induced Movement Therapy (CIMT) and Bilateral Training (BT) are two widely used neurorehabilitation approaches aimed at improving upper limb motor recovery after stroke; however, evidence comparing their effectiveness on wrist spasticity and hand function in chronic stroke patients remains limited.

This single-blinded randomized controlled trial aims to compare the effects of Constraint-Induced Movement Therapy combined with Functional Electrical Stimulation (FES) versus Bilateral Training combined with Functional Electrical Stimulation on wrist spasticity and hand function in patients with chronic stroke. A total of 94 participants diagnosed with chronic stroke will be randomly allocated into two groups. Group A will receive CIMT with FES, while Group B will receive Bilateral Training with FES. Both interventions will be administered three times per week for eight weeks.

Outcome measures will include wrist spasticity assessed using the Modified Ashworth Scale (MAS) and upper limb motor function assessed using the Fugl-Meyer Assessment for Upper Extremity (FMA-UE) and the Chedoke Arm and Hand Activity Inventory (CAHAI). Assessments will be conducted at baseline and after completion of the intervention period.

The findings of this study are expected to provide evidence on the comparative effectiveness of CIMT and Bilateral Training in improving wrist spasticity and hand function, thereby assisting clinicians in selecting optimal rehabilitation strategies for chronic stroke patients.

DETAILED DESCRIPTION:
This study is designed as a single-blinded randomized controlled trial to evaluate and compare the therapeutic effects of Constraint-Induced Movement Therapy (CIMT) and Bilateral Training (BT), both combined with Functional Electrical Stimulation (FES), on wrist spasticity and hand function in individuals with chronic stroke. Upper limb motor impairment and spasticity are major contributors to functional disability in stroke survivors, particularly in the chronic stage where spontaneous recovery is minimal and structured rehabilitation becomes essential.

Eligible participants with chronic stroke will be recruited from tertiary care hospitals and rehabilitation centers. After obtaining informed consent, participants will be randomly assigned to one of two intervention groups using a computer-generated randomization method. Outcome assessors will remain blinded to group allocation to minimize assessment bias.

Group A will receive CIMT combined with FES. CIMT will involve restraining the non-affected upper limb to encourage intensive use of the affected limb during functional and task-specific activities. Functional Electrical Stimulation will be applied to the wrist extensor muscles to facilitate muscle activation, improve motor control, and reduce spasticity.

Group B will receive Bilateral Training combined with FES. Bilateral Training will emphasize simultaneous use of both upper limbs through symmetrical and functional task-oriented activities to enhance interhemispheric coordination and promote neuroplasticity. FES parameters will remain consistent across both groups to ensure intervention standardization.

Both groups will receive therapy sessions three times per week for eight weeks, following the FITT principle. Outcome measures will be recorded at baseline and after completion of the intervention protocol. Wrist spasticity will be assessed using the Modified Ashworth Scale, while upper limb motor recovery and hand function will be evaluated using the Fugl-Meyer Assessment for Upper Extremity and the Chedoke Arm and Hand Activity Inventory.

This study aims to generate clinically relevant evidence to determine which rehabilitation approach offers superior outcomes in reducing spasticity and improving hand function in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke in chronic phase. Patients with normal cognition (MMS 21 and above) Both male and female patients will be included. Adult patients will be included. (age 18-65) Participants with spasticity score of 2 or less on MAS.

Exclusion Criteria:

* Acute and other neurological and musculoskeletal conditions e.g. Parkinson's, multiple sclerosis. Patients who do not agree to treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Change in Wrist Spasticity | 8 weeks
  Wrist spasticity will be assessed using the Modified Ashworth Scale (MAS), which grades resistance to passive movement from 0 (no increase in muscle tone) to 4 (rigid limb).

CONTACTS AND LOCATIONS:
Overall Officials: Zikra Azhar, MSPTN, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- Shadman Medical Center, Lahore, Punjab Province, Pakistan